CLINICAL TRIAL: NCT00226863
Title: Meditation and Hypnosis for Chronic Depressed Mood
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1HSA698
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2005-09-27 (Estimated); Status verified 2005-09

CONDITIONS: Long Term Depressed Mood
MeSH Terms: interventions — Meditation; Educational Status; Psychotherapy, Group; Hypnosis

INTERVENTIONS:
Behavioral: meditation plus education
Behavioral: group psychotherapy with hypnosis plus education
Behavioral: education

SUMMARY:
This study examined whether meditation or group psychotherapy including hypnosis plus education, compared to an educational control, would ameliorate long-term depressed mood.

ELIGIBILITY:
Inclusion Criteria:

* Currently meeting DSM-IV criteria for a chronic depressive disorder, with the requirement that depressive symptoms had to have lasted for at least 2 years without a remission of 2 months or more.
* Being 18 years of age or older.
* Being sufficiently proficient in English to be able to participate in group therapy.
* Being able to attend weekly meetings at Stanford.

Exclusion Criteria:

* Concurrent bipolar disorder or severe depressive disorder (this latter was determined in supervision for the SCID interviews).
* Presence or history of psychosis.
* A current primary diagnosis of panic disorder, generalized anxiety disorder, or PTSD.
* A current primary diagnosis of drug or alcohol dependency or abuse (within the last 3 months).
* Serious suicidal risk, as defined by:
* Current suicidality, i.e., beyond simple ideation (e.g., making threats or attempts; gathering means; has a plan); OR
* Serious prior attempts (bodily harm; gathered means; hospitalization).
* Has a significant medical condition that could interfere with participation in meditation/yoga.
* Current participation in psychotherapy or a meditation group.
* Has started (or changed level or type of) prescribed antidepressant medication or St. John's Wort in the previous 3 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D. Butler, Ph.D., Study Director — Stanford University; David Spiegel, M.D., Principal Investigator — Stanford University